CLINICAL TRIAL: NCT07307287
Title: SHR-A1811 Plus Pertuzumab as Neoadjuvant Therapy for Early or Locally Advanced HR-Positive HER2-Positive Breast Cancer: A Prospective, Open-Label, Phase II Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-280
Record Dates: First submitted 2025-12-02; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: SHR-A1811; HER2-Postive Breast Cancer; HR+ Breast Cancer; Early Breast Cancer; Locally Advanced Breast Cancer
Keywords: SHR-A1811; HER2-Postive Breast Cancer; HR+ Breast Cancer; Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; dalpiciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 + Pertuzumab Neoadjuvant Therapy for HER2+ HR+ Breast Cancer (Experimental): All patients to be included in the analysis must undergo Blueprint genomic profiling before neoadjuvant therapy to define luminal and non-luminal molecular subtypes. After completing four cycles of neoadjuvant therapy with ruikang-trastuzumab plus pertuzumab, response is assessed by RECIST 1.1:
  1. Patients with stable disease (SD) and luminal subtype switch to a quadruplet regimen of trastuzumab, pyrotinib, dalpiciclib, and an aromatase inhibitor for a further four cycles.
  2. Patients achieving partial or complete response (PR/CR) and luminal subtype, as well as all non-luminal patients, continue ruikang-trastuzumab plus pertuzumab for an additional 2-4 cycles, tailored to individual clinical response, before undergoing surgery
  Interventions: Drug: SHR- A1811

INTERVENTIONS:
Drug: SHR- A1811 — SHR-A1811 4.8 mg/kg and pertuzumab 420 mg are administered intravenously every 3 weeks for 4 cycles as neoadjuvant therapy. Patients with luminal subtype and stable disease (SD) then switch to trastuzumab 6 mg/kg, pyrotinib 320 mg po daily, dalpiciclib 125 mg po days 1-21 of a 28-day cycle, plus an aromatase inhibitor for 4 additional cycles. All remaining patients (PR/CR luminal or any non-luminal) continue SHR-A1811 + pertuzumab for 2-4 more cycles before surgery. Treatment continues until progression, unacceptable toxicity, or surgical resection.
  Other Names: Pyrotinib; Dalpiciclib

SUMMARY:
Breast cancer is the most common malignancy in women, with approximately 20% classified as HER2-positive. Anti-HER2 blockade (trastuzumab plus pertuzumab) combined with chemotherapy constitutes the standard neoadjuvant regimen; however, the pathological complete response (pCR) rate in the HR-positive subgroup remains only 35-40%, and platinum-containing schedules are associated with significant hematologic toxicity. Antibody-drug conjugates (ADCs) integrate targeted delivery with potent cytotoxic payloads. SHR-A1811 (ruikang-trastuzumab), a domestically developed ADC by Hengrui Pharmaceutical, is conjugated with a topoisomerase I inhibitor (mean drug-to-antibody ratio [DAR] ≈ 6). Preclinical data demonstrate that SHR-A1811 exhibits superior efficacy to trastuzumab emtansine (T-DM1) in both trastuzumab-sensitive and resistant HER2-expressing tumor models, with a manageable safety profile.

This prospective, open-label, phase II trial will enroll patients with early-stage/locally advanced HR-positive/HER2-positive breast cancer, who will receive neoadjuvant SHR-A1811 plus pertuzumab. At baseline, BluePrint gene profiling will be performed to stratify participants into luminal and non-luminal subtypes: patients with luminal subtype who achieve stable disease (SD) after 4 cycles will switch to a regimen of trastuzumab, pyrotinib, dalpiciclib, and an aromatase inhibitor for an additional 4 cycles; all other patients will continue ADC-based dual-target therapy for 2-4 further cycles, followed by surgical resection. Circulating tumor DNA (ctDNA) dynamics will be dynamically monitored at baseline, after 4 cycles of treatment, and preoperatively to evaluate early treatment sensitivity.

The primary endpoint is the pCR rate. Secondary endpoints include event-free survival (EFS), objective response rate (ORR), and safety profiles. Exploratory analyses will investigate the correlation between molecular subtypes and treatment responses, aiming to establish a chemotherapy-free, precision neoadjuvant strategy for HR-positive/HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 18-70 years at the time of informed consent.
2. Histologically confirmed invasive breast cancer, with no prior systemic anti-cancer therapy.
3. Pathologically documented HR-positive (ER ≥ 1% and/or PR ≥ 1%) and HER2-positive disease, per the 2018 ASCO-CAP guidelines: IHC 3+ or IHC 2+ with ISH ratio ≥ 2.0.
4. Clinical stage II-III (cT2-cT4 or cN+, cM0) per the 8th edition of the AJCC Cancer Staging Manual.
5. At least one measurable lesion per RECIST v1.1 criteria.
6. ECOG performance status 0-1.
7. Estimated life expectancy of ≥ 12 months.
8. Adequate organ function within 14 days prior to the first dose (without transfusion or growth factor support):

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; platelets ≥ 100 × 10⁹/L; hemoglobin (Hb) ≥ 90 g/L
   2. Albumin ≥ 3.0 g/dL; total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); alanine transaminase (ALT)/aspartate transaminase (AST) ≤ 2.5 × ULN; alkaline phosphatase (ALP) ≤ 2.5 × ULN; blood urea nitrogen (BUN) and creatinine ≤ 1.5 × ULN, or creatinine clearance (CrCl) ≥ 60 mL/min (per Cockcroft-Gault formula)
   3. Prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
   4. Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiography
   5. Fridericia-corrected QT interval (QTcF) ≤ 470 ms
9. Premenopausal women with reproductive potential must have a negative serum β-human chorionic gonadotropin (β-hCG) test within 7 days before treatment, use effective barrier contraception throughout the study period and for 6 months after the last dose, and not be breastfeeding.
10. Provision of signed written informed consent; willingness to comply with all study visits and procedures.

Exclusion Criteria:

1. Breast cancer not confirmed by histopathology.
2. Bilateral, inflammatory, or occult breast cancer.
3. Any prior anti-cancer therapy (chemotherapy, radiotherapy, targeted, endocrine, etc.); radical radiotherapy ≤ 4 weeks or palliative radiotherapy ≤ 2 weeks before first dose.
4. Concomitant anti-cancer therapy of any kind.
5. Other malignancies within 5 years (except cured basal-cell skin cancer or cervical carcinoma in situ).
6. Participation in another drug trial ≤ 4 weeks before enrolment.
7. Systemic immunosuppressive therapy (e.g., > 10 mg/day prednisone equivalent) ≤ 2 weeks before first dose (nasal/inhaled corticosteroids allowed).
8. Live or attenuated vaccines ≤ 4 weeks before first dose.
9. Major non-breast surgery ≤ 4 weeks before first dose or not fully recovered.
10. Active autoimmune disease or history of recurrent autoimmunity (e.g., autoimmune hepatitis, uveitis, colitis, hypophysitis, vasculitis, nephritis, hyper/hypothyroidism except stable hormone replacement). Controlled vitiligo, psoriasis, alopecia, insulin-dependent type 1 diabetes, or childhood asthma in complete remission allowed. Asthma requiring bronchodilators excluded.
11. Immunodeficiency (HIV positive, congenital/secondary), prior organ transplant.
12. Uncontrolled or significant cardiovascular/cerebrovascular disease, including within 6 months: NYHA III/IV heart failure, MI, stroke (except lacunar), pulmonary embolism, unstable angina, significant arrhythmia; cardiomyopathies; QTc > 470 ms (Fridericia, female), 2nd/3rd degree AV block, atrial fibrillation ≥ EHRA 2b, uncontrolled hypertension.
13. Interstitial lung disease or any moderate-severe pulmonary disorder that may interfere with drug-related lung toxicity assessment: idiopathic pulmonary fibrosis, organizing pneumonia/bronchiolitis obliterans, pulmonary embolism, severe asthma/COPD, restrictive/obstructive defects, autoimmune/connective-tissue lung involvement, prior pneumonectomy.
14. Active hepatitis B (HBsAg+ and HBV DNA ≥ 500 IU/mL), hepatitis C (anti-HCV+ and HCV RNA > ULN), cirrhosis, or severe infection requiring antibiotics/antivirals/antifungals.
15. Hereditary/acquired bleeding or thrombotic diatheses (e.g., hemophilia, coagulopathy).
16. Known hypersensitivity to study drugs or excipients.
17. Pregnant or lactating women; women of child-bearing potential with positive baseline pregnancy test or unwilling to use effective contraception throughout the study.
18. Any severe concomitant condition jeopardizing patient safety or compliance (e.g., uncontrolled hypertension, diabetes, active infection) or significant neurologic/psychiatric disorder (epilepsy, dementia) that, in the investigator's opinion, renders

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | At the time of definitive surgery, approximately 24 weeks after study entry
  Percentage of patients with no invasive cancer in the breast and axillary lymph nodes (ypT0/is ypN0) at definitive surgery.

SECONDARY OUTCOMES:
5-year Event-free survival (EFS) | 60 weeks
  5 years event-free survival after surgery
Objective response rate (ORR) | 18 weeks
  Proportion of patients achieving complete or partial response (CR + PR) by RECIST 1.1 after neoadjuvant therapy.
Safety and tolerability | From enrollment to the end of treatment at 8 weeks
  Incidence and severity of adverse events graded by CTCAE v5.0 from first dose up to 30 days after last dose.

OTHER OUTCOMES:
Exploratory biomarker analyses | 1) Tumor tissue (baseline biopsy) will be collected at baseline; 2) Peripheral blood tissue will be collected at baseline, following four cycles of treatment (each cycle is 21 days), and prior to surgery;
  1. Association between baseline molecular subtypes (luminal vs non-luminal);
  2. Cell-free tumor DNA (ctDNA) will be dynamically monitored at baseline, following four cycles of treatment, and prior to surgery;
  3. Multi-gene profiling for identifying genomic characteristics predictive of benefit from neoadjuvant SHR-A1811 plus pertuzumab in HR-positive/HER2-positive breast cancer.

IPD SHARING:
Plan to Share IPD: No